CLINICAL TRIAL: NCT01428258
Title: Phase 2 Study of Glycomacropeptide vs. Amino Acid Diet for the Management of PKU
Brief Title: Phase 2 Study of Glycomacropeptide Versus Amino Acid Diet for Management of Phenylketonuria
Acronym: PKU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-2010-0165; 1R01FD003711-01A1 (FDA)
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: Phenylketonuria
Keywords: Diet therapy; Low phenylalanine diet; Attention; Executive function
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Intervention Model Description: The study is a randomized, two-arm, crossover trial comparing the GMP diet and the AA diet in 30 subjects with PKU > 12 years of age. Subjects were randomized to start with either the GMP diet or the AA diet which they followed for 3-wk at home, followed by a 3-wk washout period when they resumed their usual AA diet, and then 3-wk of either the GMP diet or the AA diet whichever they did not consume first. Each subject served as their own control; there was no control group. We studied medical foods - either AA or GMP medical foods which are not drugs. The FDA did not require that we have an IND.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GMP Diet/GMP Medical Foods (Experimental): The experimental intervention is the GMP diet followed at home for 3-wk. In this randomized crossover study, half of subjects (n=15) were randomized to receive the GMP diet as the first arm, and half of the subjects (n=15) were randomized to receive the GMP diet as the second arm.
  Interventions: Other: AA Diet/AA Medical Foods
- AA Diet/AA Medical Foods (Active Comparator): The experimental intervention is the AA diet followed at home for 3-wk. In this randomized crossover study, half of subjects (n=15) were randomized to receive the AA diet as the first arm, and half of the subjects (n=15) were randomized to receive the AA diet as the second arm.
  Interventions: Other: GMP Diet/GMP Medical Foods

INTERVENTIONS:
Other: GMP Diet/GMP Medical Foods — The intervention consists of a low-phenylalanine (Phe) diet in combination with medical foods made with the peptide GMP supplemented with limiting indispensable amino acids, as provided by Cambrooke Therapeutics, LLC. The diet is formulated to replace the protein equivalents provided by AA medical foods with GMP medical foods, keeping other dietary components constant. The GMP dietary treatment period consists of all subjects following the GMP diet for 3-wks at home. The GMP diet intervention is administered in differing orders, GMP Diet/AA Diet or AA diet/GMP Diet.
  Other Names: GMP Medical Foods; Glytactin trademark of Cambrooke Therapeutics,LLC
  Arms: AA Diet/AA Medical Foods
Other: AA Diet/AA Medical Foods — The intervention consists of a low-Phe diet in combination with commercial AA medical foods as consumed in each subject's usual diet. A total of 15 different commercial AA medical foods were consumed by subjects in the study. The diet is formulated to provide each subject with their typical daily intake of protein equivalents from AA medical foods. The AA dietary treatment period consists of all subjects following the AA diet for 3-wks at home. The AA Diet comparator intervention is administered in differing orders, GMP Diet/AA Diet or AA diet/GMP Diet.
  Other Names: AA Medical Foods
  Arms: GMP Diet/GMP Medical Foods

SUMMARY:
For individuals with Phenylketonuria (PKU), the investigators hypothesize that glycomacropeptide will provide an acceptable form of low-phenylalanine dietary protein that will improve dietary compliance, blood phenylalanine levels, cognitive function, and ultimately quality of life compared with the usual amino acid based diet. The study is funded by the Food and Drug Administration (FDA) Office of Orphan Products Development Grants Program, R01 FD003711.

DETAILED DESCRIPTION:
Individuals with phenylketonuria (PKU) lack the enzyme phenylalanine hydroxylase that is needed to metabolize the essential amino acid phenylalanine (phe). When eating a normal diet they show an elevated level of phe in blood that is toxic to the brain. In order to prevent brain damage and cognitive impairment, individuals with PKU must follow a lifelong, low-phe diet that is restricted in natural foods and requires ingestion of a phe-free amino acid (AA) formula. Most adolescents and adults with PKU find the AA formula unpalatable and go off the diet resulting in elevated blood phe levels and neuropsychological deterioration. Glycomacropeptide (GMP), an intact protein produced during cheese making, is uniquely suited to a low-phe diet because it is the only known dietary protein that contains minimal phe. Foods and beverages made with GMP are a palatable alternative to AA formula. The long term goal is to assess the safety, efficacy and acceptability of GMP for the nutritional management of PKU. The specific aim is to conduct a randomized, two-stage, 11-wk, crossover trial comparing the GMP diet with the AA diet in 30 subjects with PKU ≥12 years of age treated since birth with a low-phe AA diet. The sites are: University of Wisconsin-Madison, Waisman Center (primary) and Harvard University, Children's Hospital Boston. Subjects will be recruited and randomized to begin the first 3-wk of the study with either a low-phe diet in which the majority of dietary protein is provided by GMP or AA medical foods and then, after a 3-wk washout with intake of their usual diet, begin the second diet for 3-wk. Dietary education will be provided in a 1-wk base period preceding initiation of each diet.

ELIGIBILITY:
Inclusion Criteria:

* Identified PKU by newborn screening; started diet treatment before 1 mo age
* Diagnosis of classical or variant PKU with documented phenylalanine level of greater than 600 umol/L at 7-10d of age
* Follows or willing to follow PKU diet and consume amino acid medical formula providing more than 50% of protein needs
* Acceptance of glycomacropeptide foods determined prior to enrollment

Exclusion Criteria:

* Females who are pregnant or planning pregnancy
* Individuals with mental deficits due to untreated or poorly controlled PKU
* Individuals with any health condition deemed to interfere with participation

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise M Ney, PhD, RD, Study Director — Professor of Nutritional Sciences, University of Wisconsin-Madison
Locations (2):
- United States (2):
  - Children's Hospital of Boston, Boston, Massachusetts
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Calcar SC, MacLeod EL, Gleason ST, Etzel MR, Clayton MK, Wolff JA, Ney DM. Improved nutritional management of phenylketonuria by using a diet containing glycomacropeptide compared with amino acids. Am J Clin Nutr. 2009 Apr;89(4):1068-77. doi: 10.3945/ajcn.2008.27280. Epub 2009 Feb 25. PMID 19244369
- [Background] Ney DM, Gleason ST, van Calcar SC, MacLeod EL, Nelson KL, Etzel MR, Rice GM, Wolff JA. Nutritional management of PKU with glycomacropeptide from cheese whey. J Inherit Metab Dis. 2009 Feb;32(1):32-9. doi: 10.1007/s10545-008-0952-4. Epub 2008 Oct 29. PMID 18956251
- [Background] Ney DM, Hull AK, van Calcar SC, Liu X, Etzel MR. Dietary glycomacropeptide supports growth and reduces the concentrations of phenylalanine in plasma and brain in a murine model of phenylketonuria. J Nutr. 2008 Feb;138(2):316-22. doi: 10.1093/jn/138.2.316. PMID 18203898
- [Background] MacLeod EL, Clayton MK, van Calcar SC, Ney DM. Breakfast with glycomacropeptide compared with amino acids suppresses plasma ghrelin levels in individuals with phenylketonuria. Mol Genet Metab. 2010 Aug;100(4):303-8. doi: 10.1016/j.ymgme.2010.04.003. Epub 2010 Apr 14. PMID 20466571
- [Background] Laclair CE, Ney DM, MacLeod EL, Etzel MR. Purification and use of glycomacropeptide for nutritional management of phenylketonuria. J Food Sci. 2009 May-Jul;74(4):E199-206. doi: 10.1111/j.1750-3841.2009.01134.x. PMID 19490325
- [Result] Ney DM, Stroup BM, Clayton MK, Murali SG, Rice GM, Rohr F, Levy HL. Glycomacropeptide for nutritional management of phenylketonuria: a randomized, controlled, crossover trial. Am J Clin Nutr. 2016 Aug;104(2):334-45. doi: 10.3945/ajcn.116.135293. Epub 2016 Jul 13. PMID 27413125
- [Result] Stroup BM, Held PK, Williams P, Clayton MK, Murali SG, Rice GM, Ney DM. Clinical relevance of the discrepancy in phenylalanine concentrations analyzed using tandem mass spectrometry compared with ion-exchange chromatography in phenylketonuria. Mol Genet Metab Rep. 2016 Jan 16;6:21-6. doi: 10.1016/j.ymgmr.2016.01.001. eCollection 2016 Mar. PMID 27014575
- [Result] Ney DM, Murali SG, Stroup BM, Nair N, Sawin EA, Rohr F, Levy HL. Metabolomic changes demonstrate reduced bioavailability of tyrosine and altered metabolism of tryptophan via the kynurenine pathway with ingestion of medical foods in phenylketonuria. Mol Genet Metab. 2017 Jun;121(2):96-103. doi: 10.1016/j.ymgme.2017.04.003. Epub 2017 Apr 6. PMID 28400091
- [Result] Stroup BM, Murali SG, Nair N, Sawin EA, Rohr F, Levy HL, Ney DM. Dietary amino acid intakes associated with a low-phenylalanine diet combined with amino acid medical foods and glycomacropeptide medical foods and neuropsychological outcomes in subjects with phenylketonuria. Data Brief. 2017 Jun 7;13:377-384. doi: 10.1016/j.dib.2017.06.004. eCollection 2017 Aug. PMID 28664173
- [Result] Stroup BM, Sawin EA, Murali SG, Binkley N, Hansen KE, Ney DM. Amino Acid Medical Foods Provide a High Dietary Acid Load and Increase Urinary Excretion of Renal Net Acid, Calcium, and Magnesium Compared with Glycomacropeptide Medical Foods in Phenylketonuria. J Nutr Metab. 2017;2017:1909101. doi: 10.1155/2017/1909101. Epub 2017 May 4. PMID 28546877
- [Result] Stroup BM, Ney DM, Murali SG, Rohr F, Gleason ST, van Calcar SC, Levy HL. Metabolomic Insights into the Nutritional Status of Adults and Adolescents with Phenylketonuria Consuming a Low-Phenylalanine Diet in Combination with Amino Acid and Glycomacropeptide Medical Foods. J Nutr Metab. 2017;2017:6859820. doi: 10.1155/2017/6859820. Epub 2017 Dec 31. PMID 29464117
- [Result] Stroup BM, Nair N, Murali SG, Broniowska K, Rohr F, Levy HL, Ney DM. Metabolomic Markers of Essential Fatty Acids, Carnitine, and Cholesterol Metabolism in Adults and Adolescents with Phenylketonuria. J Nutr. 2018 Feb 1;148(2):194-201. doi: 10.1093/jn/nxx039. PMID 29490096
- [Result] Stroup BM, Hansen KE, Krueger D, Binkley N, Ney DM. Sex differences in body composition and bone mineral density in phenylketonuria: A cross-sectional study. Mol Genet Metab Rep. 2018 Feb 3;15:30-35. doi: 10.1016/j.ymgmr.2018.01.004. eCollection 2018 Jun. PMID 30023287
- See also: National PKU Alliance — http://www.npkua.org

RESULTS

PARTICIPANT FLOW:
Groups:
- GMP Diet-AA Diet: In this randomized crossover study, half of subjects will be assigned to an arm that consists of the the GMP diet followed by the AA diet referred to as the Glycomacropeptide (GMP) diet given first intervention.
  Glycomacropeptide (GMP) diet given first: The intervention compares a new low-phenylalanine (phe) dietary therapy for PKU, a diet containing foods and beverages made from GMP using Glytactin provided by Cambrooke Foods LLC, with the usual amino acid (AA) low-phe dietary therapy. PKU subjects in the GMP Diet-AA Diet Arm will follow the GMP diet that will replace all of the dietary protein equivalents provided by AA formula with foods and beverages made from GMP for 3 weeks followed by a 3 wk wash out period. They will then follow the usual AA diet for 3 weeks. Each dietary treatment period will maintain constant intake of total protein and phe and last for 3 weeks in subjects living at home.
- AA Diet - GMP Diet: In this randomized crossover study, half of subjects will be assigned to an arm that consists of the AA diet followed by the GMP diet referred to as the Amino Acid (AA) Diet given first intervention.
  Amino Acid (AA) Diet Given First: The intervention compares the usual amino acid (AA) low-phenylalanine (phe) dietary therapy with a new dietary therapy for PKU, a low-phe diet containing foods and beverages made from glycomacropeptide (GMP). PKU subjects in the AA Diet-GMP Diet Arm will follow their usual AA diet for 3 weeks followed by a 3 wk wash out period. They will then replace all of the protein equivalents provided in their diet by AA formula with foods and beverages made from GMP using Glytactin as provided by Cambrooke Foods, LLC. Each dietary treatment period will maintain constant intake of total protein and phe and last for 3 weeks in subjects living at home.
Period: Intervention 1
Arm/Group | GMP Diet-AA Diet | AA Diet - GMP Diet
Started | 17 | 15
Completed | 15 | 15
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Intervention 2
Arm/Group | GMP Diet-AA Diet | AA Diet - GMP Diet
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GMP Diet-AA Diet | AA Diet - GMP Diet | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 5
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 28 [15 to 56] | 28 [15 to 56] | 28 [15 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 3 | 10 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in the Plasma Phenylalanine Concentration of PKU Subjects Fed the Glycomacropeptide Diet Compared With the Change When Fed the Amino Acid Diet
Description: Plasma will be collected at each base week and after 3 weeks on each of the dietary treatments, glycomacropeptide and amino acid, following an overnight fast. Plasma phenylalanine concentration (along with the complete profile of free amino acids) will be determined with an amino acid analyzer in the Wisconsin State Lab of Hygiene. Statistical analysis to determine the significance of the change in plasma phe concentration when comparing the 2 diets will consist of ANCOVA with covariates for baseline Phe and dietary Phe intake. The change in plasma Phe concentration from day 22 (final) to day 1 (baseline) was determined after adjusting for baseline Phe level and dietary Phe intake.
Time Frame: baseline to day 22 on each diet
Measure: Mean (Standard Error); unit: micro moles per liter plasma
Groups:
- GMP Diet/GMP Medical Foods: All subjects received the Glycomacropeptide (GMP) diet either in the first or second period. The intervention consists of a low-Phe diet in combination with medical foods made from glycomacropeptide, a low-Phe whey protein.
- AA Diet/AA Medical Foods: All subjects received the Amino Acid (AA) Diet in either the first or second period. The intervention consists of a low-Phe diet in combination with each subject's usual AA medical formula.
Arm/Group | GMP Diet/GMP Medical Foods | AA Diet/AA Medical Foods
Number analyzed (Participants) | 30 | 30
micro moles per liter plasma | 62 (40) | -85 (40)
Statistical Analysis 1: Comparison: GMP Diet/GMP Medical Foods vs AA Diet/AA Medical Foods; Test type: Superiority or Other; p = 0.0008, ANCOVA; Mean Difference (Net) = -147, Standard Error of Mean 39
Statistical Analysis 2: Comparison: GMP Diet/GMP Medical Foods; Test type: Other; p = 0.136, ANCOVA
Statistical Analysis 3: Comparison: AA Diet/AA Medical Foods; Test type: Other; p = 0.044, ANCOVA

2. Secondary Outcome: Dietary Compliance
Description: Compliance with the glycomacropeptide and amino acid dietary treatments will be assessed by comparison of the intake of medical food in grams of protein from medical food per day based on subject completion of 3-day food records prior to the final study visit on day 22. Statistical analysis for a dietary treatment effect will consist of ANOVA.
Time Frame: 3 week dietary treatment
Measure: Mean (Standard Error); unit: g protein from MF/kg/day
Groups:
- GMP Diet: All subjects received the Glycomacropeptide (GMP) diet either in the first or second period. The intervention consists of a low-Phe diet in combination with medical foods made from glycomacropeptide, a low-Phe whey protein.
Arm/Group | GMP Diet | AA Diet/AA Medical Foods
Number analyzed (Participants) | 30 | 30
g protein from MF/kg/day | 0.74 (0.04) | 0.76 (0.05)
Statistical Analysis 1: Comparison: GMP Diet vs AA Diet/AA Medical Foods; Test type: Other; p = 0.576, ANOVA

3. Secondary Outcome: Executive Function Assessed by BRIEF
Description: Completion of a standardized test, the Behavior Rating Inventory of Executive Function (BRIEF), by each subject for the GMP diet and the AA diet. Values are T-scores which have a mean of 50 points and a SD of 10 points. A T score of <50 is considered within the normative range. Data are analyzed with a paired t-test.
Time Frame: day 22 of each dietary treatment
Measure: Mean (Standard Error); unit: T score
Groups:
- GMP Diet/GMP Medical Foods: The intervention followed as the first or second treatment consists of a low-Phe diet in combination with medical foods made from glycomacropeptide .
- AA Diet/AA Medical Foods: The intervention followed as the first or second treatment consists of a low-Phe diet in combination with each subjects usual AA medical foods.
Arm/Group | GMP Diet/GMP Medical Foods | AA Diet/AA Medical Foods
Number analyzed (Participants) | 30 | 30
T score | 49.0 (1.8) | 48.8 (2.1)
Statistical Analysis 1: Comparison: GMP Diet/GMP Medical Foods vs AA Diet/AA Medical Foods; Test type: Other; p = 0.902, t-test, 2 sided

4. Secondary Outcome: Vitamin D (25-OH) Plasma Concentration at Day 22
Description: Vitamin D was measured as a measure of the capacity for calcium absorption. Higher levels of plasma vitamin D are consistent with higher calcium absorption.
Time Frame: day 22 of each dietary treatment
Measure: Mean (Standard Error); unit: ng per ml
Arm/Group | GMP Diet/GMP Medical Foods | AA Diet/AA Medical Foods
Number analyzed (Participants) | 30 | 30
ng per ml | 33.8 (1.70) | 33.6 (1.52)
Statistical Analysis 1: Comparison: GMP Diet/GMP Medical Foods vs AA Diet/AA Medical Foods; Test type: Other; p = 0.797, t-test, 2 sided

5. Secondary Outcome: Comparison of Phe Concentrations in Plasma With Concentrations in Dried Blood Spots
Description: Concentrations of Phe in plasma and in dried blood spots collected simultaneously by subjects will be compared using 2 methodologies, regardless of intervention. At each of the 4 study visits (baseline and final for each dietary treatment): 1) venipuncture was used to collect blood and plasma was isolated and analyzed for Phe with ion exchange chromatography and 2) subjects were asked right after the venipuncture to spot their blood on filter paper for analysis of Phe with tandem mass spectroscopy (MS/MS). The discrepancy in Phe concentrations with these 2 methods was compared for each sample pair using Bland-Altman statistical analysis. Each subject should have had 4 sample pairs, 29 x 4 = 116, but we ended up with only 110 sample pairs, as explained below.
Time Frame: 4 times total, 2 per treatment
Population: Analysis of sample pairs is required to determine the discrepancy in Phe levels with the 2 methods. Each subject should have had 4 sample pairs, 29 x 4 = 116, but we ended up with only 110 sample pairs. The explanation for the difference is that several subjects did not provide dried blood spots because research staff forgot to obtain them.
Measure: Mean (Standard Error); unit: micro moles per liter
Groups:
- Phe Concentration in Plasma, Ion Exchange Chromatography: Blood was collected by venipuncture at 3 to 4 time points, plasma was isolated and the concentration of Phe was determined by ion exchange chromatography.
- Phe Concentration in Dried Blood Spots, Tandem Mass Spec: Subjects spotted their blood on filter paper at the same time as plasma was obtained at 3 or 4 time periods, dried blood spots were obtained, and analyzed for Phe concentration using tandem mass spectrometry.
Arm/Group | Phe Concentration in Plasma, Ion Exchange Chromatography | Phe Concentration in Dried Blood Spots, Tandem Mass Spec
Number analyzed (Participants) | 29 | 29
micro moles per liter | 731 (32) | 514 (23)
Statistical Analysis 1: Comparison: Phe Concentration in Plasma, Ion Exchange Chromatography vs Phe Concentration in Dried Blood Spots, Tandem Mass Spec; Test type: Other; p = 0.0001, ANOVA

6. Secondary Outcome: Bone-specific Alkaline Phosphatase (BSAP) Plasma Concentration at Day 22
Description: Plasma concentration of BSAP was determined as a measure of bone turnover.
Time Frame: day 22 of each dietary treatment
Population: Samples were not obtained from 4 subjects due to a collection error by research staff. Thus the sample size is reduced from 30 to 26.
Measure: Mean (Standard Error); unit: micro gram per liter
Groups:
- GMP Diet/GMP Medical Foods: The intervention followed as the first or second treatment consists of a low-Phe diet in combination with medical foods made with glycomacropeptide.
Arm/Group | GMP Diet/GMP Medical Foods | AA Diet/AA Medical Foods
Number analyzed (Participants) | 26 | 26
micro gram per liter | 17.0 (2.1) | 17.0 (2.2)

7. Secondary Outcome: N-terminal Telopeptide (NTX) Plasma Concentration at Day 22
Description: Plasma concentration of NTX was determined as a measure of bone resorption; higher levels indicate greater bone breakdown
Time Frame: day 22 of each dietary treatment
Population: Samples were not obtained from 3 subjects due to a collection error by research staff. Thus the sample size is reduced from 30 to 27.
Measure: Mean (Standard Error); unit: nmol per liter bone collagen equivalents
Groups:
- GMP Diet/GMP Medical Foods: The intervention administered as the first or second dietary treatment consists of a low-Phe diet in combination with medical foods made with glycomacropeptide.
- AA Diet/AA Medical Foods: The intervention administered as the first or second dietary treatment consists of a low-Phe diet in combination with each subjects usual AA medical foods.
Arm/Group | GMP Diet/GMP Medical Foods | AA Diet/AA Medical Foods
Number analyzed (Participants) | 27 | 27
nmol per liter bone collagen equivalents | 17.5 (0.66) | 17.1 (0.65)

8. Other Pre Specified Outcome: Bone Mineral Density Determined by Dual-energy X-ray Absorptiometry (DXA) Scan
Description: Subjects will have a single DXA test to assess bone mineral density of the lumbar spine and total body during the first dietary treatment that they are randomly assigned to start with.
Time Frame: once during first 3 week dietary treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For each subject, adverse events were monitored for each of the 3-wk treatment periods for each diet.
Arm/Group | GMP Diet/GMP Medical Foods | AA Diet/AA Medical Foods
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/30

LIMITATIONS AND CAVEATS:
The trial was completed as planned with an adequate number of subjects and there were no limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No